CLINICAL TRIAL: NCT04634617
Title: Pelvic Floor Dysfunction and Quality of Life in Uterine Cancer Survivors
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2018-0242; NCI-2019-08260 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0242 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-11-09; First posted 2020-11-18 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Endometrial Carcinoma; Malignant Uterine Neoplasm; Uterine Corpus Cancer; Uterine Corpus Sarcoma
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaires): Patients complete questionnaires over 45-60 minutes consisting of demographic, treatment, lifestyle, disease, and comorbidity questions, as well as multiple study instruments assessing quality of life as it pertains to common toxicities of uterine cancer treatment.
  Interventions: Other: Questionnaire Administration

INTERVENTIONS:
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This trial studies pelvic floor dysfunction and quality of life in uterine cancer survivors. Using questionnaires may help researchers learn more about the sexual function and quality of life in uterine cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate and compare the prevalence of pelvic floor dysfunction in uterine cancer survivors by modality of treatment and to compare with a control group with no history of cancer using the Pelvic Floor Distress Inventory (PFDI).

SECONDARY OBJECTIVES:

I. To compare the degree of sexual dysfunction in uterine cancer survivors by modality of treatment using the Female Sexual Function Index (FSFI) as a continuous measure, and to compare to a non-cancer control group.

II. To compare the long term quality of life (QoL) (using the FSFI, the Pelvic Floor Impact Questionnaire [PFIQ], Functional Assessment of Cancer Therapy-Endometrial Cancer [FACT-En], Brief Pain Inventory [BPI], Alzheimer's Disease Assessment Scale [ADAS]/Cancer Rehabilitation Evaluation System for Research [CARES] dating scale and Menopausal survey) of patients who were treated with surgery and radiotherapy versus surgery alone (with or without chemotherapy), and to compare to a control group with no history of cancer.

III. To evaluate associations between dose volume parameters of organs at risk and pelvic floor symptoms using the PFIQ and PFDI.

IV. To evaluate associations between the radiation and surgical technique and quality of life (including pelvic symptoms and sexual function using the FSFI, PFIQ, PFDI, and FACT-En).

OUTLINE:

Patients complete questionnaires over 45-60 minutes consisting of demographic, treatment, lifestyle, disease, and comorbidity questions, as well as multiple study instruments assessing quality of life as it pertains to common toxicities of uterine cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with uterine cancer (including endometrial and uterine carcinoma or sarcoma) treated with surgery +/- radiation at MD Anderson between 2006 and 2017

  * Eligible surgeries include laparoscopic or robotic assisted abdominal total hysterectomy, total abdominal hysterectomy, and vaginal hysterectomy with or without pelvic node dissection, with or without omentectomy or omental biopsies
  * In addition, patients must have had all WITH bilateral-salpingo-oophorectomy (BSO), either during their surgery or in a previous or subsequent (within 3 months of endometrial cancer diagnosis) surgery
* Patients have had at least one year of follow-up
* Patients have not had any recurrence of disease
* Patients must be able to complete the survey of their own volition
* Patients must be able to read and speak English fluently
* CONTROL GROUP: Patients have never been diagnosed with any cancer other than non-melanomatous skin cancers
* CONTROL GROUP: Patient has undergone hysterectomy/BSO for benign reasons between 2006 and 2017
* CONTROL GROUP: Patients must be able to complete the survey of their own volition
* CONTROL GROUP: Patients must be able to speak and read English fluently

Exclusion Criteria:

* Patients with cancer recurrence, as this will affect their current quality of life
* Patients with additional pelvic surgery at the time of their hysterectomy (for example pelvic exenteration, urostomy placement, etc.)
* Patients with a secondary primary cancer (including cervical cancer), as this will affect their current quality of life. Patients may have either squamous cell or basal cell carcinoma of the skin
* Neurocognitive deficits that render patients unable to complete the survey on their own
* Patients who have not yet had removal of their bilateral ovaries
* Preoperative radiotherapy prior to hysterectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with uterine cancer treated with surgery +/- radiation at MD Anderson between 2006 and 2017 and patients who have never been diagnosed with any cancer other than non-melanomatous skin cancers and have undergone hysterectomy/bilateral-salpingo-oophorectomy (BSO) for benign reasons between 2006 and 2017
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2027-04-11 (Estimated); Study Completion 2027-04-11 (Estimated)

PRIMARY OUTCOMES:
Pelvic floor distress (PFD) | Up to 1 year
  Measured by the Pelvic Floor Distress Inventory-20. Descriptive statistics (i.e. frequencies, percentages, medians, ranges, means, standard deviations, measures of skewness and kurtosis), including 95% confidence intervals (CIs) will be computed for the measures derived by study cohort. Prevalence estimates along with exact 95% CIs will be computed. Logistic regression analysis will be used to assess the odds of PFD for treatment cohorts relative to the cohort of patient controls.

CONTACTS AND LOCATIONS:
Overall Officials: Lilie L Lin, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org